CLINICAL TRIAL: NCT06130436
Title: Application of Perioperative Remote Ischemic Conditioning in Patients Undergoing Hepatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRIC
Record Dates: First submitted 2023-11-02; First posted 2023-11-14 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2023-10

CONDITIONS: Hepatic Hemangioma; Liver Cancer; Hepatolithiasis; Hepatectomy
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, patient-assessor blinded, sham-controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sham-Remote Ischemic Conditioning (Sham Comparator): Sham remote ischemic conditioning (Sham-RIC) is applied in the perioperative using an automated Sham-RIC device.
  Interventions: Device: Sham-Remote Ischemic Conditioning
- Remote Ischemic Conditioning Once Daily (Active Comparator): Remote ischemic conditioning (RIC) is applied in the perioperative using an automated RIC device once daily.
  Interventions: Device: Remote Ischemic Conditioning Once Daily
- Remote Ischemic Conditioning Twice Daily (Active Comparator): Remote ischemic conditioning (RIC) is applied in the perioperative using an automated RIC device twice daily.
  Interventions: Device: Remote Ischemic Conditioning Twice Daily

INTERVENTIONS:
Device: Sham-Remote Ischemic Conditioning — Sham-Remote Ischemic Conditioning (at the time points of 30 min before anesthesia, 30 min after surgery, the morning of the postoperative day 1, the afternoon of the postoperative day 1, the morning of the postoperative day 2, the afternoon of the postoperative day 2): Three cycles (30 minutes), each consisting of five minutes of cuff inflation followed by five minutes with a deflated cuff, but the cuff pressure will be 0 mmHg.
  Arms: Sham-Remote Ischemic Conditioning
Device: Remote Ischemic Conditioning Once Daily — Remote Ischemic Conditioning (at the time points of 30 min before anesthesia, the morning of the postoperative day 1, the morning of the postoperative day 2): Three cycles (30 minutes), each consisting of five minutes of cuff inflation followed by five minutes with a deflated cuff. The cuff pressure will be 200 mmHg.
  Sham-Remote Ischemic Conditioning (at the time points of 30 min after surgery, the afternoon of the postoperative day 1, the afternoon of the postoperative day 2): Three cycles (30 minutes), each consisting of five minutes of cuff inflation followed by five minutes with a deflated cuff, but the cuff pressure will be 0 mmHg.
  Arms: Remote Ischemic Conditioning Once Daily
Device: Remote Ischemic Conditioning Twice Daily — Remote Ischemic Conditioning (at the time points of 30 min before anesthesia, 30 min after surgery, the morning of the postoperative day 1, the afternoon of the postoperative day 1, the morning of the postoperative day 2, the afternoon of the postoperative day 2): Three cycles (30 minutes), each consisting of five minutes of cuff inflation followed by five minutes with a deflated cuff. The cuff pressure will be 200 mmHg.
  Arms: Remote Ischemic Conditioning Twice Daily

SUMMARY:
Our primary aim is to investigate whether perioperative remote ischemic conditioning (PRIC) as an adjunctive treatment can improve postoperative recovery in patients undergoing hepatectomy as an adjunct to standard treatment.

DETAILED DESCRIPTION:
Remote Ischemic Conditioning (RIC) can be applied as repeated short-lasting ischemia in a distant tissue that results in protection against subsequent long-lasting ischemic injury in the target organ. This protection can be applied prior to or during a prolonged ischemic event as remote ischemic pre-conditioning (RIPreC) and per-conditioning (RIPerC), respectively, or immediate after reperfusion as remote ischemic post-conditioning (RIPostC).

RIC is a non-pharmacologic and non-invasive treatment without noticeable discomfort, commonly achieved by inflation of a blood pressure cuff to induce 5-minute cycles of limb ischemia alternating with 5 minutes of reperfusion. However, whether perioperative remote ischemic conditioning (PRIC) can improve postoperative recovery in patients undergoing hepatectomy has never been investigated in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hepatectomy under general anesthesia
* American Society of Anesthesiology (ASA) grade of II ~ III
* Male and female patients, age 25 to 75 years
* New York Heart Association (NYHA) grade of I ~ III

Exclusion Criteria:

* Patients with limb deformity or peripheral vascular disease affecting upper limb function
* Patients with a medical history of nervous system, immune system and mental illness
* Patients who have received hepatectomy in the past, have important organ diseases or have undergone surgical treatment recently
* Patients who have recently used anti-inflammatory analgesics, anticoagulants, hormone drugs, immunosuppressants, and ATP-sensitive K-channel blockers (KATP)
* Preoperative severe renal insufficiency (serum creatinine > 442 umol/L, with or without serum potassium > 6.5 mmol/L, or the clinician-recognized need for renal replacement therapy), liver insufficiency (Child-Pugh grade C)
* Patients and/or their family members refuse to participate in the program

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2023-11-02 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-08-09 (Actual)

PRIMARY OUTCOMES:
Alanine aminotransferase (ALT) | 7 days
  The levels of ALT in perioperative period

SECONDARY OUTCOMES:
Aspartate aminotransferase (AST) | 7 days
  The levels of AST in perioperative period
Total bilirubin (TBIL) | 7 days
  The levels of TBIL in perioperative period
International normalized ratio (INR) | 7 days
  The levels of INR in perioperative period
Albumin (ALB) | 7 days
  The levels of ALB in perioperative period
Tumor necrosis factor-α (TNF-α) | 7 days
  The levels of TNF-α in perioperative period
Malondialdehyde (MDA) | 7 days
  The levels of MDA in perioperative period
Heme oxygenase-1 (HO-1) | 7 days
  The levels of HO-1 in perioperative period
Nuclear Factor-κB (NF-κB) | 7 days
  The levels of NF-κB in perioperative period
High mobility group box1 (HMGB1) | 7 days
  The levels of HMGB1 in perioperative period
Platelet | 7 days
  The levels of platelet in perioperative period
White blood cell (WBC) | 7 days
  The levels of WBC in perioperative period
Neutrophil granulocyte percentage | 7 days
  The levels of neutrophil granulocyte percentage in perioperative period
Time to gastrointestinal tolerance | 7 days
  Gastrointestinal tolerance was defined as transanal or stoma defecation and oral dietary tolerance.
Prolonged postoperative ileus | 7 days
  Prolonged postoperative ileus was diagnosed if patients met two or more of the following conditions on or after postoperative day 4: inability to tolerate the oral diet over the past 24 h, nausea or vomiting, without flatus over the past 24 h, abdominal distension or radiological evidence of intestinal distension without mechanical intestinal obstruction.
Rate of postoperative complications | 30 days
  The postoperative complications were recorded using the Clavien-Dindo classification system and included: nausea or vomiting, abdominal distension, anastomotic leakage, new pulmonary infection, poor wound healing, cognitive dysfunction, unplanned reoperation, and 30-day readmission rate.

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, ph.D, Study Chair — The Second Affiliated Hospital, Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital, Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data for this study is available from the sponsor on reasonable request through email.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 3 months and ending 2 years following article publication.
Access Criteria: To gain access data requestors will need to sign a data processing agreement.

REFERENCES:
- [Derived] Tian C, Tian H, Li W, Chen J, Guo Q, Duan G, Huang H. Effects of Remote Ischemic Conditioning on Postoperative Recovery After Hepatectomy: A Randomised Controlled Trial. Liver Int. 2025 Mar;45(3):e70041. doi: 10.1111/liv.70041. PMID 39982031